CLINICAL TRIAL: NCT00074568
Title: Scleroderma Family Registry and DNA Repository
Brief Title: Scleroderma Registry
Acronym: Registry
Status: Completed | Type: Observational
Sponsor: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Collaborators: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Sponsor
Other Study IDs: NIAMS-108; N01AR002251-000 (NIH); NO1-AR-0-2251
Record Dates: First submitted 2003-12-16; First posted 2003-12-17 (Estimated); Last update posted 2022-09-27 (Actual); Status verified 2022-09

CONDITIONS: Systemic Sclerosis; Scleroderma
Keywords: Genetic Study; Transmission Dysequilibrium Testing; Genome Wide Scan; Family Study
MeSH Terms: conditions — Scleroderma, Systemic; Scleroderma, Diffuse

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, Plasma, DNA
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Patients with scleroderma and their family members (parents, brothers, and sisters)
- 2: Healthy volunteers with no autoimmune disease and without a first-degree relative with a systemic autoimmune disease

SUMMARY:
Scleroderma is likely caused by a combination of factors, including an external trigger (infection or other exposure) and a genetic predisposition. The Scleroderma Registry will conduct genetic analyses for disease-related genes in patients with scleroderma and their family members (parents, brothers, and sisters).

DETAILED DESCRIPTION:
Scleroderma refers to a group of diseases that involve the abnormal growth of connective tissue, which supports the skin and internal organs. Scleroderma can affect the skin, making it hard and tight; it can also damage the blood vessels and internal organs such as the heart, lungs, and kidneys. Estimates for the number of people in the United States with the systemic (body-wide) form of scleroderma range from 40,000 to 165,000. The number of people with all scleroderma-related disorders is between 250,000 and 992,500.

Researchers believe that several factors interact to produce scleroderma, including abnormal immune activity, potential environmental triggers, and genetic makeup. Scleroderma is not passed on from parents to child, but certain genes may make a person more likely to develop the disease. The goals of this project are to identify the genes that influence disease susceptibility and expression in systemic scleroderma and to establish a repository of DNA, plasma, and serum samples from single case scleroderma families, multicase families, and healthy unrelated volunteers for the use of researchers interested in studying this disease.

Participants in the Registry will have a phone interview regarding disease characteristics and family history. Participants will be sent a blood kit to get a blood sample drawn locally for shipment to the Registry lab. Blood samples will be made available (anonymously) for studies by researchers around the country. In some cases, participants will be asked to sign a release of medical information so that medical records can be obtained to verify the diagnosis.

As of May 2009, this study is no longer enrolling family members.

ELIGIBILITY:
Inclusion Criteria

* Diagnosis of systemic sclerosis or family members of patients with systemic sclerosis

Or

* Healthy volunteer with no autoimmune disease and without a first-degree relative with a systemic autoimmune disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with Systemic Sclerosis or family member of patients with systemic sclerosis
  or
  Healthy volunteer with no autoimmune disease and without a first degree relative with a systemic autoimmune disease.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Actual)
Dates: Start 2000-09; Primary Completion 2022-01 (Actual); Study Completion 2022-01 (Actual)

PRIMARY OUTCOMES:
Establish National registry of Scleroderma as resource for scleroderma scientific community | ongoing

CONTACTS AND LOCATIONS:
Overall Officials: Maureen D. Mayes, MD, MPH, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- University of Texas - Houston Medical School, Houston, Texas, United States

REFERENCES:
- [Background] Mayes MD, Giannini EH, Pachman LM, Buyon JP, Fleckman P. Connective tissue disease registries. Arthritis Rheum. 1997 Sep;40(9):1556-9. doi: 10.1002/art.1780400903. No abstract available. PMID 9324008
- [Background] Mayes MD. The establishment and utility of a population-based registry to understand the epidemiology of systemic sclerosis. Curr Rheumatol Rep. 2000 Dec;2(6):512-6. doi: 10.1007/s11926-000-0029-3. PMID 11123106
- [Background] Mayes MD. Scleroderma epidemiology. Rheum Dis Clin North Am. 2003 May;29(2):239-54. doi: 10.1016/s0889-857x(03)00022-x. PMID 12841293